CLINICAL TRIAL: NCT00723242
Title: The Role of Dendritic Cells in Hepatitis C Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Professor Nikolai V. Naoumov
Purpose: Basic Science
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — Ribavirin

INTERVENTIONS:
Drug: Viraferon-peg and Rebetol

SUMMARY:
The role of the dendritic cells, the most potent antigen presenting cells, in the establishment of chronic hepatitis C is not established. The study aims to define whether the dendritic cells are affected by the hepatitis C virus and whether that bears an impact on the antiviral immune response they generate. The hypothesis is explored by investigating a group of patients prior to and after the initiation of standard treatment for hepatitis C with pegylated Interferon and Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* anti-HCV positive
* HCV RNA positive

Exclusion Criteria:

* contraindications for antiviral treatment
* concurrent chronic viral infections

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Basic science research (immunology of hepatitis C)in hepatitis c patients receiving established, standard antiviral treatment (pegylated Interferon+Ribavirin)

CONTACTS AND LOCATIONS:
Locations (1):
- University College Hospital, London, United Kingdom